CLINICAL TRIAL: NCT02931929
Title: MITIGATE-NeoBOMB1: A Phase I/IIa Study to Evaluate Safety, Biodistribution, Dosimetry+Preliminary Diagnostic Performance of 68Ga-NeoBOMB1 in Pat. With Advanced TKI-treated GIST Using Positron-emission Tomography/Computer Tomography (PET/CT)
Brief Title: MITIGATE-NeoBOM: A Study to Evaluate 68Ga- NeoBOMB1 in Patients With Advanced TKI-treated GIST Using PET/CT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Irene Virgolini, Univ.-Prof. Dr. med., Medical University Innsbruck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MITIGATE-NeoBOMB1
Record Dates: First submitted 2016-09-29; First posted 2016-10-13 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-NeoBOMB1 (Other): 68Ga-NeoBOMB1, 2-vial kit for radiolabelling. I.v. Administration after radiolabelling
  Interventions: Drug: 68Ga-NeoBOMB1, 2-vial kit

INTERVENTIONS:
Drug: 68Ga-NeoBOMB1, 2-vial kit — intravenous application of a radiopharmaceutical for Positron Emission tomography (PET)
  Other Names: NeoBOMB1

SUMMARY:
Tyrosine-kinase Inhibitors (TKI) resistance in gastrointestinal stromal tumours (GIST) is a common problem after prolonged treatment periods. The main objectives of this monocentric diagnostic Phase I/IIa study are safety and tolerability, pharmacokinetics and dosimetry of 68Ga-NeoBomb1 in GIST patients. The rationale behind this study is to improve diagnostic accuracy in GIST via positron-emission tomography/computer tomography (PET-CT) with a focus on TKI-resistant subtypes. Better detection, classification and definition of lesion extent are expected from the use of 68Ga-NeoBOMB1.

DETAILED DESCRIPTION:
Rationale of the design:

This is a monocentric diagnostic Phase I/IIa study. Due to the very limited number of patients and the rare nature of the disease the study was designed as a combination of phases I and IIa.

The main objectives of such an early phase clinical trial are safety and tolerability, pharmacokinetics and (in the case of radiopharmaceuticals) dosimetry aspects. For the first 6 patients, the focus of the study will be on safety, tolerability and pharmacokinetics. Therefore, both TKI-resistant and TKI-sensitive GIST patients will be included. As resistant patients are typically in 2nd- or 3rd-line TKI treatment prone to substantial side effects and potentially suffer from a greater extent of disease, the study design includes a limited number of non-resistant GIST patients to address a possible bias regarding tolerability and side effects profile of 68Ga-NeoBOMB1.

After 6 included patients an interim analysis of safety and pharmacokinetic data including PBPK modelling and dosimetry calculation will be performed. Thereby it will be decided, whether the data generation is sufficient for a final calculation of dosimetry, if so pharmacological and dosimetric aspects can be omitted in the last 6 patients, reducing the burden for these patients considerably (less number of scans, no blood and urine sampling). This analysis will also reveal the optimal time window for PET/CT imaging.

After the establishment of these baseline findings, the second part of the study will emphasize the assessment of imaging data towards targeting properties of the GRP(gastrin releasing peptide)-receptor-specific radiopharmaceutical 68Ga-NeoBOMB1 as proof of the molecular imaging principle. In this phase only patients with confirmed GRPR receptor expression via Immunohistochemistry will be included. Nonetheless, safety and tolerability still remain a primary objectives in this part of the study.

As there are no preclinical indications that the GRP receptor status of TKI resistance is variable, all objectives should be met including targeting properties of 68Ga-NeoBOMB1 also in non-resistant patients. Nonetheless, changes in GRP-receptor expression under treatment pressure may still exist. Therefore in both phases a minimum of 50% of the patients have to show resistance to TKI treatment, where therapeutic option are extremely limited. This will allow providing data in patients that will most likely benefit most from an improved target characterisation and GRPR targeting therapy approaches.

Study conduct:

Within 28 days after the patient's positive evaluation and written informed consent, the imaging study will be performed. During the study, patients will be shortly hospitalised. These pre-planned hospitalisations for study purposes will not be considered as (serious) adverse events. The radiopharmaceutical will be administered to the patient directly at the imaging system (PET-CT).

In the first phase of the trial including the first six patients a series of dynamic scans between 0 and 45 min and static whole-body PET images at 1, 2 and 3-4h will be obtained to determine pharmacokinetics and absorbed doses to normal organs and to tumorous lesions. Blood samples drawn concomitantly at the time of imaging will be collected to estimate residence times in blood and to derive the bone marrow absorbed dose (max. 10 samples during the hospitalisation). Urine will be collected to determine the bladder wall and kidney absorbed doses. Regions of interest for critical organs and tumour lesions will be drawn using the acquired images resulting in time-activity curves with quantitative fractions of administered activity. Residence times of radioactivity from this analysis will be calculated. All dosimetric calculations will be performed by feeding the residence times as well as blood and urine activities into an appropriate software program (OLINDA/EXAM).

The second phase is in principle conducted in the same way, if interim analysis returns sufficient data for dosimetry and pharmacokinetics, PET images will be reduced to 2 whole body scans within the optimal time window and blood and urine sampling can be omitted.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures
* Patients with histologically confirmed advanced GIST
* Previous or current TKI treatment
* A minimum of 50% of patients showing either 1st-, 2nd- or 3rd-line TKI-resistance documented either through RECIST 1.1 criteria, Choi-criteria or FDG-CT/PET and showing presence of at least one surgically untreatable primary or metastasis confirmed with either 18F-FDG PET/CT or structural imaging (CT, MRI) and a minimum of 25% non-resistant patients.
* Karnofsky performance status > 70%
* Age > 21 years.
* Participating men must use a single barrier method for contraception for 1 month after completion of the trial starting at the day of application of 68Ga-NeoBOMB1.
* Women of childbearing age must use two highly effective methods of contraception during the trial and 6 months after its completion if not in menopause (defined as onset of menopause without menstruation for over 1 year) or after hysterectomy.

The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly effective:

* Oral hormonal contraception ('pill') (as far as its efficacy is not expected to be impaired during the trial, e.g. with IMPs that cause vomiting and diarrhoea, adequate safety cannot be assumed)
* Dermal hormonal contraception
* Vaginal hormonal contraception (NuvaRing®)
* Contraceptive plaster
* Long-acting injectable contraceptives
* Implants that release progesterone (Implanon®)
* Tubal ligation (female sterilisation)
* Intrauterine devices that release hormones (hormone spiral)
* Double barrier methods
* This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).
* The regulations for contraception are derived from Guideline ICH E8 Chapter 3.2.2.1 Selection of subjects together with ICH M3 Note 4 - Confirmed GRPR expression in tumour lesion(s) by immunohistochemistry or PCR (phase IIa only)

Exclusion Criteria:

* Renal insufficiency with an eGFR < 45 ml/min/1.72m2 or intolerance to any constituents of intravenous CT-contrast agents, preventing their administration (in cases without an available recent and sufficient contrast-enhanced CT examination)
* Higher than grade 2 hematotoxicity (CTC > 2)
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and without evidence of recurrence for 5 years
* Participation in any other investigational trial within 30 days of study entry with potential interactions regarding the study drugs or the underlying disease
* Pregnancy, breast-feeding
* Patients with concurrent illnesses that might preclude study completion or interfere with study results
* Patients with bladder outflow obstruction or unmanageable urinary incontinence
* Known or expected hypersensitivity, to 68Gallium, Bombesin or to any of the excipients of NeoBOMB1.
* Any condition that precludes raised arms position for prolonged imaging purposes.
* Prior administration of a radiopharmaceutical within a period corresponding to 8 half-lives of the radionuclide used on such radiopharmaceutical.
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product.
* Subjects with any kind of dependency on the investigator or employed by the sponsor or investigator
* Subjects held in an institution by legal or official order

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | day 12-20 after administration
  Patients will undergo physical examinations, ECG, blood pressure measurements as well as analysis of blood biochemistry (haemoglobin, haematocrit, RBC count, WBC count, absolute neutrophil count, differential WBC count (neutrophils, eosinophils, basophils, lymphocytes, monocytes [%]), platelets), haematology (glucose, urea, creatinine, eGFR (calculated), bilirubin, Na, K, Cl, Ca, GOT [ASAT], GPT [ALAT], γGT, pancreas lipase and amylase, ALP, LDH, CK, CRP, serum albumin), coagulation parameters (Quick, INR, aPTT, fibrinogen) and semi-quantitative urine analysis (leukocytes, nitrite, erythrocytes, pH, protein). These measurements and assessments will be repeated during and after the application of 68Ga-NeoBOMB1. Prior to the study inclusion, prior to application of 68Ga-NeoBOMB1 and during the second follow-up a potential pregnancy will be assessed. The presence and severity of adverse events will be judged and reported according to CTCAE v4.03.
Organ and compartment dosimetry data, human pharmacokinetics of 68Ga-NeoBOMB1 and identification of potentially dose-limiting organs | 3-4 hours after administration
  Pharmacokinetic data will be acquired by measuring 68Ga-NeoBOMB1 distribution over time through successive dynamic/semi-dynamic/static PET scans. Time activity curves will be generated to determine relative distribution among and doses for all relevant organs and compartments [% of injected radioactivity in MBq] through a physiology-based pharmacokinetic modelling approach (OLINDA/EXAM).
  To gather more information, successive blood and urine sampling will also be used to provide blood activity and excretion information and estimate bloodpool/bone marrow doses.
Preliminary targeting properties of 68Ga-NeoBOMB1 in advanced, GRP positive GIST tumours as assessed by SUV | 3-4 hours after administration
  GIST lesion tracer accumulation will be assessed visually and measured as relative signal intensity (compared to blood pool activity, SUV) for known lesions.

SECONDARY OUTCOMES:
Targeting properties in comparison with standard imaging modalities such as FDG-PET or MRI as assessed by sensitivity and specificity | 3-4 hours after administration
  The lesion demarcation from 68Ga-NeoBOMB1-PET will be compared to contrast-enhanced computed tomography and FDG-PET (if available).
Qualitative comparison of targeting properties of 68Ga-NeoBOMB1 in resistant vs non-resistant tumour lesions in patients undergoing TKI Treatment as assessed by presence of tracer uptake and SUV | 3-4 hours after administration
  Relative lesion growth tendency (as calculated from comparing current and previous CT scans) will be correlated to their respective tracer uptake (SUV).
Identification of target tissue and improved target volume definition for potential locoregional treatment (RFA or external beam) | 3-4 hours after administration
  A comparison will be made whether 68Ga-NeoBOMB1-PET could offer additional information for a potential local therapy such as radiofrequency ablation (RFA) or external beam radiation as determined by definition of lesion amount and extent.
  Therapeutic interventions will not be part of the current study
To extrapolate absorbed tumour doses for potential application of 177Lu NeoBOMB1 (in first 6 patients) | 3-4 hours after administration
  Estimation of tumour and organ/compartment doses will be performed by means of a physiology-based pharmacokinetic modelling to assess the potential feasibility of a therapeutic approach of 177Lu-NeoBOMB1

CONTACTS AND LOCATIONS:
Overall Officials: Irene Virgolini, Univ-Prof.Dr, Principal Investigator — Head of department of nuclear medicine
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No